CLINICAL TRIAL: NCT02431780
Title: A Multi-centre, Randomised, Controlled, Clinical Investigation of a Standalone Decision Support Algorithm for Neonatal Seizure Recognition
Brief Title: A Multicentre Clinical Investigation of a Decision Support Algorithm for Neonatal Seizure Detection
Acronym: ANSeR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Collaborators: University College, London (Other); Wellcome Trust (Other)
Responsible Party: Principal Investigator, Professor Geraldine Boylan, Professor, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GB01/14UCC
Record Dates: First submitted 2014-11-14; First posted 2015-05-01 (Estimated); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Seizures; Brain Diseases; Central Nervous System Diseases; Epilepsy; Nervous System Diseases; Neurologic Manifestations
Keywords: Neonatal Seizures; Decision Support Algorithm; EEG
MeSH Terms: conditions — Seizures; Brain Diseases; Central Nervous System Diseases; Epilepsy; Nervous System Diseases; Neurologic Manifestations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- non ANSeR Software System (No Intervention): Routine clinical EEG monitoring
- ANSeR Software System (Experimental): The intended use of the ANSeR Software System is to provide a real time decision support tool to assist in the diagnosis of seizures in neonates (between 36 weeks and 44 weeks corrected age) and to provide a review tool for EEG and seizure analysis. ANSeR is intended to provide a reliable, effective, objective and intuitive means of identifying seizures
  Interventions: Device: ANSeR Software System

INTERVENTIONS:
Device: ANSeR Software System — ANSeR Software System a stand alone, software medical device for Neonatal seizure decision support tool
  Arms: ANSeR Software System

SUMMARY:
The ANSeR Clinical Investigation is a multi-centre, randomised, controlled, clinical investigation of a standalone decision support Algorithm for Neonatal Seizure Recognition, the ANSER Software system.

DETAILED DESCRIPTION:
This will be an open, two arm, parallel group, randomised, controlled investigation of the ANSeR Software System as a stand-alone neonatal seizure recognition decision support tool. Term neonates requiring EEG monitoring will be stratified by recruiting site and then randomised to receive either EEG monitoring with the ANSeR Software System or EEG monitoring without the ANSeR Software System.

It is proposed that the rate of true detections (sensitivity) of investigation personnel using the ANSeR Software System in clinical practice will be at least 25% higher than that of investigation personnel not using the ANSeR Software System in routine clinical practice. In addition we expect the specificity of investigation personnel using the ANSeR Software System to be no worse than 10% less than that of investigation personnel not using the ANSeR Software System. This should result in more appropriate and timely use of antiepileptic drugs (AED).

Randomisation Immediately following enrolment in the investigation, each participant will be randomly assigned to receive either EEG monitoring with the ANSeR Software System or without the ANSeR Software System. Randomisation will be stratified by recruiting site with a 1:1 allocation ratio to each group. Block randomisation with varying block sizes will be used and the randomisation and allocation will be performed centrally using a web-based electronic system.

Blinding As this is an investigation of a medical device (software), the investigation personnel will be aware of which group the participant is assigned to. The expert panel who are the diagnostic reference standard will be blinded to group allocation. The biostatistician will also be blinded to group allocation during the analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

* Neonates 36 weeks - 44 weeks corrected gestational age in whom EEG monitoring is indicated because they are deemed to be

  * at high risk of seizures or
  * are experiencing seizures

Exclusion Criteria:

* • No parental/guardian consent

Ages: 36 Weeks to 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 264 (Actual)
Dates: Start 2015-02-12 (Actual); Primary Completion 2017-02-07 (Actual); Study Completion 2017-02-07 (Actual)

PRIMARY OUTCOMES:
The Seizure Detection Rate for all Neonates enrolled in the investigation arm compared to Seizure Detection Rate for all Neonates in the control arm. | 12-18 months
  The rate of true seizure detection (sensitivity), as recorded on a Seizure Record form, 25% superior in the investigation arm compared to the control group (usual clinical practice). The Expert Committee will be used as the diagnostic reference standard.
The False Detections per hour (sensitivity) for all Neonates enrolled in the investigation arm compared to the False Detection Rate for all Neonates in the control arm. | 12-18 months
  The False Detections per hour (specificity), as recorded on a Seizure Record form, 10% superior in the investigation arm compared to the control group (usual clinical practice). The Expert Committee will be used as the diagnostic reference standard.

SECONDARY OUTCOMES:
Seizure burden (min) for all Neonates enrolled in the investigation arm compared to Seizure burden (min) for all Neonates in the control arm. | 12-18 months
  To quantify seizure burden (min) in the investigation arm and control arm.
Number of Neonates administered Anti-epileptic drug (AED) in the investigation arm compared to Number of Neonates administered Anti-epileptic drug (AED) in the control arm. | 12-18 months

CONTACTS AND LOCATIONS:
Overall Officials: Janet Rennie, Doctor, Principal Investigator — University College London Hospitals; Geraldine Boylan, PhD, Principal Investigator — University College Cork, Cork, Ireland
Locations (8):
- Ireland (2):
  - Cork University Maternity Hospital, Wilton, Cork
  - Rotunda Maternity Hospital, Dublin
- University Medical Centre Utrecht, Wilhelmina Children's Hospital, Utrecht, Netherlands
- Karolinska Institutet and University Hospital, Huddinge, Stockholm County, Sweden
- United Kingdom (4):
  - Barts and the London NHS Trust,, London
  - The London and Homerton Hospital, London
  - University College London Hospitals NHS Foundation Trust, London
  - Great Ormond Street Hospital, London

REFERENCES:
- [Result] Pavel AM, Rennie JM, de Vries LS, Blennow M, Foran A, Shah DK, Pressler RM, Kapellou O, Dempsey EM, Mathieson SR, Pavlidis E, van Huffelen AC, Livingstone V, Toet MC, Weeke LC, Finder M, Mitra S, Murray DM, Marnane WP, Boylan GB. A machine-learning algorithm for neonatal seizure recognition: a multicentre, randomised, controlled trial. Lancet Child Adolesc Health. 2020 Oct;4(10):740-749. doi: 10.1016/S2352-4642(20)30239-X. Epub 2020 Aug 27. PMID 32861271
- [Result] Pavel AM, O'Toole JM, Proietti J, Livingstone V, Mitra S, Marnane WP, Finder M, Dempsey EM, Murray DM, Boylan GB; ANSeR Consortium. Machine learning for the early prediction of infants with electrographic seizures in neonatal hypoxic-ischemic encephalopathy. Epilepsia. 2023 Feb;64(2):456-468. doi: 10.1111/epi.17468. Epub 2022 Dec 20. PMID 36398397
- [Result] Pavel AM, Mathieson SR, Livingstone V, O'Toole JM, Pressler RM, de Vries LS, Rennie JM, Mitra S, Dempsey EM, Murray DM, Marnane WP, Boylan GB; ANSeR Consortium. Heart rate variability analysis for the prediction of EEG grade in infants with hypoxic ischaemic encephalopathy within the first 12 h of birth. Front Pediatr. 2023 Jan 4;10:1016211. doi: 10.3389/fped.2022.1016211. eCollection 2022. PMID 36683815
- [Result] Pavel AM, Rennie JM, de Vries LS, Blennow M, Foran A, Shah DK, Pressler RM, Kapellou O, Dempsey EM, Mathieson SR, Pavlidis E, Weeke LC, Livingstone V, Murray DM, Marnane WP, Boylan GB. Neonatal Seizure Management: Is the Timing of Treatment Critical? J Pediatr. 2022 Apr;243:61-68.e2. doi: 10.1016/j.jpeds.2021.09.058. Epub 2021 Oct 7. PMID 34626667
- See also: ANSeR Study Research Group — http://anserstudy.com/